## Effects of Simethicone and Multilac Baby in Infantile Colic

| Doctor Information | | |
|---|---|---|
| Doctor | | |
| Date | | |
| Patient Data | | |
| General Patient Data | | |
| Patient Initials | | |
| Gender: | male | female |
| Date of birth: | | |
| Delivery type: | Normal | Ceasarian section |
| Birth in pregnancy week: | | |
| Weight at time of birth: | | |
| Breast feeding: Formula feeding: | yes | no |
| romula reeding. | yes | no |
| Antibiotics therapies: | yes | no |
| Details of antibiotics therapy: | | |
| D /G 1: 1: | | |
| Pro-/Synbiotics | yes | no |
| Details of Pro-/Syn-Therapy | | |
| Primary Diagnostics (before treatment start) | | |
| Days of crying during last 3 weeks? | | |
| Average duration of crying? | | |
| Number of crying phases per day? Can the child be calmed during crying? | 1/05 | no |
| Can the child be calified during crying: | yes | no |
| Bloated belly? | yes | no |
| Retracted legs? | yes | no |
| Red face? | yes | no |
| Problems to fall asleep? | yes | no |
| Short (<30 min) sleeping periodes during the day? | yes | no |
| Short (<16h) total sleeping time per day? | yes | no |
| Number of sleeping periodes per day? | | |
| Comments | | |
| Comments | | |